CLINICAL TRIAL: NCT02271997
Title: Optimizing Iron Suppletion After Roux-en-Y Gastric Bypass
Acronym: Ironsuppletion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ironsuppletion
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous fumarate; ferrous gluconate; ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ferrous fumarate (Active Comparator): 40 patients receive ferrous fumarate 3 times a day 200mg
  Interventions: Drug: Ferrous fumarate
- Ferrous gluconate (Active Comparator): 40 patients receive ferrous gluconate 2 times a day 695 mg
  Interventions: Drug: Ferrous gluconate
- Iron(III)carboxymaltose (Active Comparator): 40 patients receive a single intravenous shot of ferinject
  Interventions: Drug: Iron(III)carboxymaltose

INTERVENTIONS:
Drug: Ferrous fumarate — treatment with ferrous fumarate during 1 year and 6,12,26 and 52 weeks after starting treatment iron spectrum will be measured
  Arms: Ferrous fumarate
Drug: Ferrous gluconate — treatment with ferrous gluconate during 1 year and 6,12,26 and 52 weeks after starting treatment iron spectrum will be measured
  Other Names: Losferron
  Arms: Ferrous gluconate
Drug: Iron(III)carboxymaltose — treatment with Iron(III)carboxymaltose and 6,12,26 and 52 weeks after starting treatment iron spectrum will be measured
  Other Names: Ferinject
  Arms: Iron(III)carboxymaltose

SUMMARY:
Multicentre randomized controlled trial to evaluate the optimal treatment for patients who developed an iron deficiency after Roux-en-Y Gastric bypass.

DETAILED DESCRIPTION:
Morbid obesity is worldwide a still growing problem. The number of bariatric procedures are still increasing with 9000 bariatric operations in 2009. The golden standard is the Roux-en-Y Gastric bypass (RYGB). The RYGB ensures an excess weight loss of 60-70% in our hospital.

Unfortunately vitamin and mineral deficiencies are a consequence from RYGB. Iron deficiency occurs in 14-66% in the first two years after surgery. Worldwide there are three most used options of treatment for this: treatment with ferrous fumarate, ferrous gluconate and intravenous injection of Ferinject.

Our goal is to determine which treatment is the most effective to normalize ferritin values in the blood and which treatment is the most cost-effective one after a RYGB.

ELIGIBILITY:
Inclusion Criteria:

* all women who underwent a Roux-en-Y gastric bypass and developed an iron deficiency postoperatively (ferritin<20microgram/L)

Exclusion Criteria:

* iron deficiency peroperative, blood transfusions during study period, iron containing nutritional supplements except the standard multivitamins after bariatric surgery, decreased renal failure, excessive blood loss due to menstruation, anemia not caused by iron deficiency, accumulation of iron, hypersensitivity for noe of the medicinal products, psychiatric illness, pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
normal value serum ferritin | 1 year
  1 year after initiating therapy

SECONDARY OUTCOMES:
patients preference for oral or intravenous therapy | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - OLVG West/ Sint Lucas Andreas Ziekenhuis, Amsterdam, North Holland
  - Rijnstate hospital, Arnhem
  - Rose Kruis Ziekenhuis, Beverwijk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schijns W, Boerboom A, de Bruyn Kops M, de Raaff C, van Wagensveld B, Berends FJ, Janssen IMC, van Laarhoven CJHM, de Boer H, Aarts EO. A randomized controlled trial comparing oral and intravenous iron supplementation after Roux-en-Y gastric bypass surgery. Clin Nutr. 2020 Dec;39(12):3779-3785. doi: 10.1016/j.clnu.2020.04.010. Epub 2020 Apr 21. PMID 32402684